CLINICAL TRIAL: NCT01209546
Title: Study of the Effect of FLUTTER VRP1 in Patients With Bronchiectasis.
Brief Title: Study of the Effect of FLUTTER® VRP1 (PEP and Oscillating High Frequency).
Acronym: FLUTTER®VRP1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The protocol finished.
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ada Clarice Gastaldi, Professor Ada Clarice Gastaldi, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: USP 2010-2
Record Dates: First submitted 2010-07-12; First posted 2010-09-27 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2010-09

CONDITIONS: Bronchiectasis
Keywords: Bronchiectasis; Pulmonary function; Respiratory muscle strength; Respiratory secretions
MeSH Terms: conditions — Bronchiectasis | interventions — Control Groups; Population Groups; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Flutter group (Active Comparator): In Flutter group the exercise used the Flutter ®VRP1 (VarioRaw SA, Switzerland).
  Interventions: Other: Flutter group
- PEP group (Active Comparator): In PEP group the exercise used the Flutter ®VRP1 (VarioRaw SA, Switzerland) without the steel ball inside, with the closure of so many holes as necessary to produce a positive expiratory pressure equivalent to pressure achieved by patients during the performance with the ball in the Flutter®VRP1.
  Interventions: Other: PEP group
- control group (Placebo Comparator): In placebo patients were assessed as pulmonary function, respiratory muscle strength and transport properties of respiratory secretions
  Interventions: Other: control group
- Group Sham (Sham Comparator): Exercise with Flutter®VRP1 without the ball inside
  Interventions: Other: Group Sham

INTERVENTIONS:
Other: control group — In placebo patients were assessed and were not subjected to any respiratory physical therapy technique.
  Other Names: group without therapy
  Arms: control group
Other: Flutter group — Patients have done exercise sessions with Flutter ®VRP1 for 30 minutes daily in a randomized, crossover, with four weeks of treatment with a therapy, a week of wash-out followed by four more weeks with the other modality (PEP).
  Other Names: Futter VRP1 device without modification
  Arms: Flutter group
Other: PEP group — Patients have done exercise sessions with Flutter® VRP1 without the steel ball inside, with the closure of so many holes as necessary to produce a positive expiratory pressure equivalent to pressure achieved by patients during the performance with the ball in the Flutter®VRP1 for 30 minutes daily in a randomized, crossover, with four weeks of treatment with a therapy, a week of wash-out followed by four more weeks with the other modality (Flutter®VRP1).
  Other Names: Flutter VRP1 without the ball inside
  Arms: PEP group
Other: Group Sham — Patients have done exercise sessions with Flutter ®VRP1 for 30 minutes without the ball inside daily in a randomized, crossover, with four weeks of treatment with a therapy, a week of wash-out followed by four more weeks with the other modality (PEP)
  Arms: Group Sham

SUMMARY:
The research sought to assess the effects of Flutter ® VRP1 in patients with bronchiectasis.

DETAILED DESCRIPTION:
Bronchiectasis is an airway disease with many etiologies characterized pathologically by the abnormal permanent dilatation of bronchi, caused mainly by the perpetuation of inflammatory processes induced by frequent episodes of bacterial infections, with consequent change in the ciliated epithelial lining and compromising the effectiveness of mucociliary clearance that can favor the hypersecretive state found in these patients.

In addition to drug therapy or surgical treatment, patients with bronchiectasis also have physiotherapy, which is an important part in treatment. The patients present impaired mucus transport, and can enjoy the benefits provided by respiratory therapy, which features intended to increase the removal of airway secretions and thus reduce the obstruction to improve ventilation and oxygenation.

One of the instruments commonly used in respiratory therapy is the Flutter ® VRP1 (VarioRaw SA, Switzerland), which is a simple equipment, small, similar to a pipe that combines two techniques: positive expiratory pressure (PEP) and high-frequency oscillations.

Some previous studies have shown beneficial effects after use of this device in patients with bronchiectasis. However, it is unclear whether the mechanism of action is related to the combination of PEP and the techniques of high frequency oscillation, or just one of those components.

ELIGIBILITY:
Inclusion Criteria:

* Non Cystic Fibrosis Bronchiectasis
* Amount of secretion sufficient for analysis
* Capable of fulfilling the experimental protocol

Exclusion Criteria:

* Acute pulmonary disease
* Presence of any respiratory infection in the last four weeks

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2008-01 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The Effect of FLUTTER VRP1 on respiratory mucus transport | five years
  30 patients with bronchiectasis will receive sessions with the Flutter®VRP1 or PEP for 30 minutes daily in a randomized, crossover study. Weekly secretion samples will be collected and evaluated for mucociliary relative transport velocity(RTV), displacement in a simulated cough machine(SCM) and contact angle measurement(CAM).

CONTACTS AND LOCATIONS:
Overall Officials: Ada C. Gastaldi, doctor, Study Chair — University of Sao Paulo
Locations (1):
- Faculty of Medicine of Ribeirão Preto, University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Result] App EM, Kieselmann R, Reinhardt D, Lindemann H, Dasgupta B, King M, Brand P. Sputum rheology changes in cystic fibrosis lung disease following two different types of physiotherapy: flutter vs autogenic drainage. Chest. 1998 Jul;114(1):171-7. doi: 10.1378/chest.114.1.171. PMID 9674466
- [Result] Fahy JV, Schuster A, Ueki I, Boushey HA, Nadel JA. Mucus hypersecretion in bronchiectasis. The role of neutrophil proteases. Am Rev Respir Dis. 1992 Dec;146(6):1430-3. doi: 10.1164/ajrccm/146.6.1430. PMID 1280928
- [Result] Thompson CS, Harrison S, Ashley J, Day K, Smith DL. Randomised crossover study of the Flutter device and the active cycle of breathing technique in non-cystic fibrosis bronchiectasis. Thorax. 2002 May;57(5):446-8. doi: 10.1136/thorax.57.5.446. PMID 11978924
- [Derived] Tambascio J, de Souza HCD, Martinez R, Baddini-Martinez JA, Barnes PJ, Gastaldi AC. Effects of an Airway Clearance Device on Inflammation, Bacteriology, and Mucus Transport in Bronchiectasis. Respir Care. 2017 Aug;62(8):1067-1074. doi: 10.4187/respcare.05214. PMID 28733314
- See also: University of São Paulo link — http://www.fmrp.usp.br